CLINICAL TRIAL: NCT04215302
Title: Prediction Accuracy for Langeal Mask Unique TM Size in Melayu Pediatric Population According to Weight Meissurement
Brief Title: Prediction Accuracy for Langeal Mask Unique TM Size in Pediatric Patient
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Christopher Kapuangan, MD, Indonesia University
Other Study IDs: IndonesiaUAnes053
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: General Anaesthesia
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- laryngeal mask size: laryngeal mask size determines according to weight measurement
  Interventions: Device: laryngeal mask

INTERVENTIONS:
Device: laryngeal mask — the size of laryngeal mask given to the patient was based on patient's weight measurement

SUMMARY:
the study aimed to know the accuracy for laryngeal mask unique TM size to Malay pediatric race according to weight measurement recommended by manufacturer

DETAILED DESCRIPTION:
sixty-six pediatric subjects aged between 1 - 10 years old underwent general anesthesia using laryngeal mask Unique TM. Laryngeal mask inserted using the size based on subject's weight. Effectivity was confirmed if there is no air sound from patient's mouth, airway seal pressure ≥20 cmH2O, maximum inspiration pressure was ≤ 20 cmH2O, difference in expiration and inspiration tidal volume less than 5%, and there is no cuff appear in mouth.

ELIGIBILITY:
Inclusion Criteria:

* aged 1 -10 years old
* Malay race
* scheduled for general anesthesia procedure with laryngeal mask

Exclusion Criteria:

- disagree to be included in the study

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric population aged 1 - 10 years old underwent general anesthesia procedure with laryngeal mask airway device
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
successful insertion of laryngeal mask | 3 minutes
  observe the sign of successful insertion of laryngeal mask

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kapuangan, MD, Principal Investigator — Indonesia University
Locations (1):
- Indonesia University, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Michalek P, Donaldson W, Vobrubova E, Hakl M. Complications Associated with the Use of Supraglottic Airway Devices in Perioperative Medicine. Biomed Res Int. 2015;2015:746560. doi: 10.1155/2015/746560. Epub 2015 Dec 13. PMID 26783527
- [Result] Takahoko K, Iwasaki H, Sasakawa T, Suzuki A, Matsumoto H, Iwasaki H. Unilateral hypoglossal nerve palsy after use of the laryngeal mask airway supreme. Case Rep Anesthesiol. 2014;2014:369563. doi: 10.1155/2014/369563. Epub 2014 Aug 31. PMID 25254120
- [Result] Brain AI, Howard D. Lingual nerve injury associated with laryngeal mask use. Anaesthesia. 1998 Jul;53(7):713-4. doi: 10.1046/j.1365-2044.1998.537d-az0584d.x. No abstract available. PMID 9771185
- [Result] King C, Street MK. Twelfth cranial nerve paralysis following use of a laryngeal mask airway. Anaesthesia. 1994 Sep;49(9):786-7. doi: 10.1111/j.1365-2044.1994.tb04452.x. No abstract available. PMID 7978135
- [Result] Lowinger D, Benjamin B, Gadd L. Recurrent laryngeal nerve injury caused by a laryngeal mask airway. Anaesth Intensive Care. 1999 Apr;27(2):202-5. doi: 10.1177/0310057X9902700214. PMID 10212721
- [Result] Wynn JM, Jones KL. Tongue cyanosis after laryngeal mask airway insertion. Anesthesiology. 1994 Jun;80(6):1403. No abstract available. PMID 8010489
- [Result] van Zundert TC, Brimacombe JR, Ferson DZ, Bacon DR, Wilkinson DJ. Archie Brain: celebrating 30 years of development in laryngeal mask airways. Anaesthesia. 2012 Dec;67(12):1375-85. doi: 10.1111/anae.12003.x. PMID 23130725